CLINICAL TRIAL: NCT00855166
Title: A 24-week,Multi-centre,Int.,Double-blind,Rand.,Parallel-group,Plac.-Controlled,Phase III Study With a 78-week Ext.Per. to Evaluate the Effect of Dapagliflozin in Combination With Metformin on Body Weight in Subjects With Type2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: Evaluation of the Effect of Dapagliflozin in Combination With Metformin on Body Weight in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1690C00012
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Dapagliflozin; Metformin; Type 2 diabetes; body weight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight | interventions — dapagliflozin; Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Dapagliflozin 10 mg plus Metformin
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Sitagliptin
- B (Placebo Comparator): Placebo plus Metformin
  Interventions: Drug: Metformin; Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablet oral 10 mg total daily dose once daily 102 weeks
  Arms: A
Drug: Metformin — Tablet oral 1500 - 2500 mg total daily dose 1-3 times a day104 weeks
Drug: Sitagliptin — Tablet oral 100 mg total daily dose once daily rescue medication
Drug: Placebo — Matching placebo for dapagliflozin, tablet, oral, once daily, 102 weeks
  Arms: B

SUMMARY:
This study is being carried out to see if dapagliflozin in addition to metformin decreases body weight and if so, how it compares with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Ongoing treatment with metformin on a stable dose of ≥1500 mg/day for at least 12 weeks prior to enrolment
* Inadequate glycemic control, defined as HbA1c ≥6.5% and ≤8.5%
* ≥30 years for males
* ≥55 years for females

Exclusion Criteria:

* Type 1 Diabetes
* Body weight change >5% within 3 months prior to enrolment
* Renal and liver impairment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bolinder, MD, PhD, Principal Investigator — Dept of Endocrinology, Metabolism and Diabetes Karolinska University Hospital Huddinge Karolinska Institutet 141 86 Stockholm Sweden
Locations (21):
- Bulgaria (2):
  - Research Site, Blagoevgrad
  - Research Site, Sofia
- Czechia (5):
  - Research Site, Beroun
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Semily
  - Research Site, Slaný
- Hungary (5):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Kecskemét
  - Research Site, Tát
- Poland (3):
  - Research Site, Elblag
  - Research Site, Krakow
  - Research Site, Torun
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Jarfalla
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- [Derived] Bolinder J, Ljunggren O, Johansson L, Wilding J, Langkilde AM, Sjostrom CD, Sugg J, Parikh S. Dapagliflozin maintains glycaemic control while reducing weight and body fat mass over 2 years in patients with type 2 diabetes mellitus inadequately controlled on metformin. Diabetes Obes Metab. 2014 Feb;16(2):159-69. doi: 10.1111/dom.12189. Epub 2013 Aug 29. PMID 23906445
- [Derived] Ljunggren O, Bolinder J, Johansson L, Wilding J, Langkilde AM, Sjostrom CD, Sugg J, Parikh S. Dapagliflozin has no effect on markers of bone formation and resorption or bone mineral density in patients with inadequately controlled type 2 diabetes mellitus on metformin. Diabetes Obes Metab. 2012 Nov;14(11):990-9. doi: 10.1111/j.1463-1326.2012.01630.x. Epub 2012 Jun 29. PMID 22651373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 13 Feb 2009. Last participant completed 24 week period: 03 Jun 2010. 314 participants were enrolled, 182 were randomized in 40 centers in 5 European countries. Men aged 30-75 years and women aged 55-75 years with inadequate glycemic control (HbA1c 6.5% to 8.5%), BMI of at least 25 kg/sqm and body weight <= 120 kg.
Pre-assignment Details: During a placebo lead-in period, participants were counselled on dietary and life-style modifications. The metformin dose was adjusted to open label 1500 mg/day, 2000 mg/day or 2500 mg/day. Neither gender should exceed 60% of the total number of randomized participants.
Groups:
- Placebo Plus Metformin: Placebo oral once daily plus metformin over 24 weeks
- Dapagliflozin Plus Metformin: Dapagliflozin 10 mg oral once daily plus metformin over 24 weeks
Period: Overall Study
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Started | 91 | 91 (Of the 91 randomized participants only 89 were included in the full analysis set.)
Completed | 86 | 83
Not Completed | 5 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Poor/non-compliance | 2 | 0
Not completed — Administrative reasons by sponsor | 1 | 0
Not completed — Subject no longer meets study criteria | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin | Total
Number analyzed (Participants) | 91 | 89 | 180
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (6.82) | 60.6 (8.16) | 60.7 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 51 | 49 | 100
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 91 | 89 | 180
Body Weight [Mean (Standard Deviation); unit: Kilogram] | 90.91 (13.716) | 92.06 (14.128) | 91.48 (13.894)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.68 (3.890) | 32.06 (3.887) | 31.87 (3.882)
Glycosylated hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.16 (0.531) | 7.19 (0.443) | 7.17 (0.489)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: Milligram per deciliter] | 149.60 (25.086) | 148.01 (24.650) | 148.82 (24.815)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in Total Body Weight
Description: To evaluate the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin on total body weight after 24 weeks of oral administration of double-blind treatment.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 91 | 89
kg | -0.88 (0.2746) [-1.43 to -0.34] | -2.96 (0.2766) [-3.51 to -2.41]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided); with treatment group and stratum (gender) as effects and baseline value as covariate; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-2.84 to -1.31], Standard Error of Mean 0.3885

2. Secondary Outcome: Adjusted Mean Change in Waist Circumference
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 24 weeks of double-blind treatment on waist circumference.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 91 | 89
cm | -0.99 (0.4349) [-1.84 to -0.13] | -2.51 (0.4388) [-3.38 to -1.64]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0143, ANCOVA — Significant at alpha=0.05 (2-sided). Results of key secondary endpoints are interpreted using Hochberg's method; with treatment group and stratum (gender) as effects and baseline value as covariate; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-2.74 to -0.31], Standard Error of Mean 0.6162

3. Secondary Outcome: Adjusted Mean Change in Body Fat Mass
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 24 weeks of double-blind treatment on total body fat mass measured by dual energy X-ray absorptiometry.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 79 | 82
kg | -0.74 (0.2670) [-1.27 to -0.22] | -2.22 (0.2626) [-2.74 to -1.70]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided). Results of key secondary endpoints are interpreted using Hochberg's method; with treatment group and stratum (gender) as effects and baseline value as covariate; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-2.22 to -0.74], Standard Error of Mean 0.3731

4. Secondary Outcome: Proportion of Participants With Body Weight Decrease ≥5%
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 24 weeks of double-blind treatment on body weight decrease ≥5%. Least Squares Mean represents the percent of participants adjusted for body weight baseline value.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 91 | 89
Percentage of participants | 4.3 [0.1 to 8.6] | 30.6 [21.1 to 40.2]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Significant at alpha=0.05 (2-sided). Results of key secondary endpoints are interpreted using Hochberg's method; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value and stratum (gender); Risk Difference (RD) = 26.3, 95% CI 2-sided [15.9 to 36.7], Standard Error of Mean 5.309

5. Other Pre Specified Outcome: Adjusted Percent Change in Bone Mineral Density (BMD) at Lumbar Spine (L1-4)
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 102 weeks of double-blind treatment on Bone Mineral Density at lumbar spine (L1-4) as measured by Dual Energy X-ray Absorptiometry.
Time Frame: Baseline to Week 102
Population: Safety Analysis Set (all participants who received at least one dose of double-blind study medication)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Placebo Plus Metformin: Placebo oral once daily plus metformin over 102 weeks
- Dapagliflozin Plus Metformin: Dapagliflozin 10 mg oral once daily plus metformin over 102 weeks
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 71 | 68
Percent | 0.47 [-0.32 to 1.27] | 0.69 [-0.19 to 1.57]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.7013, Mixed Models Analysis — Exploratory. Model including fixed categorical effects of treatment, week, treatment-by-week interaction, gender and rescue medication as well as continuous fixed covariates of baseline measurement and baseline measurement-by-week interaction; Percent change in BMD from baseline to week 102 evaluated via longitudinal repeated measures analysis using direct likelihood; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.89 to 1.34], Standard Error of Mean 0.5652 — Natural logarithms of baseline and week 102 values were used

6. Other Pre Specified Outcome: Adjusted Percent Change in Bone Mineral Density (BMD) at Femoral Neck
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 102 weeks of double-blind treatment on Bone Mineral Density at femoral neck as measured by Dual Energy X-ray Absorptiometry.
Time Frame: Baseline to Week 102
Population: Safety Analysis Set (all participants who received at least one dose of double-blind study medication)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 71 | 68
Percent | 0.09 [-0.83 to 1.01] | -0.85 [-1.85 to 0.16]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.1521, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-2.21 to 0.35], Standard Error of Mean 0.6473 — Natural logarithms of baseline and week 102 values were used

7. Other Pre Specified Outcome: Adjusted Percent Change in Bone Mineral Density (BMD) at Total Hip
Description: To assess the effect of dapagliflozin 10 mg daily in combination with metformin compared to placebo in combination with metformin after 102 weeks of double-blind treatment on Bone Mineral Density at total hip as measured by Dual Energy X-ray Absorptiometry.
Time Frame: Baseline to Week 102
Population: Safety Analysis Set (all participants who received at least one dose of double-blind study medication)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Number analyzed (Participants) | 71 | 68
Percent | -0.37 [-1.00 to 0.26] | -0.82 [-1.52 to -0.12]
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Dapagliflozin Plus Metformin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.3105, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.32 to 0.43], Standard Error of Mean 0.4428 — Natural logarithms of baseline and week 102 values were used

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Placebo Plus Metformin | Dapagliflozin Plus Metformin
Serious Adverse Events (participants affected / at risk) | 1/91 | 6/91
Other Adverse Events (participants affected / at risk) | 9/91 | 7/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin (N=91) | Dapagliflozin Plus Metformin (N=91)
Pneumonia (Infections and infestations) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Oesophageal varices hemorrhage (Gastrointestinal disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin (N=91) | Dapagliflozin Plus Metformin (N=91)
Nasopharyngitis (Infections and infestations) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1

LIMITATIONS AND CAVEATS:
For participants who did not complete 24 weeks, last observation carried forward (LOCF) was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.